CLINICAL TRIAL: NCT05667818
Title: An Open-label, Balanced, Randomized, Two Treatment, Two Sequence, Two Period, Two Way Crossover, Single Oral Dose Comparative Pharmacokinetic Study of Amlodipine Besylate Controlled-release Tablets, EQ 5mg Base of Overseas Pharmaceuticals Ltd., China and Norvasc®(Amlodipine Besylate) Tablets, 5mg of Pfizer Laboratories Div. Pfizer Inc., in Normal, Healthy, Adult, Human Subjects Under Fasting Conditions
Brief Title: An Comparative Pharmacokinetic Study of Amlodipine Besylate Controlled-release Tablets,China in Normal, Healthy, Adult, Human Subjects Under Fasting Conditions
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Overseas Pharmaceuticals, Ltd. (Industry)
Collaborators: Guangzhou Health Start Pharmaceutical Techology Co.,Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: YYKQ-202210-2
Record Dates: First submitted 2022-12-09; First posted 2022-12-29 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2022-12

CONDITIONS: Hypertension
Keywords: Hypertension; Healthy Volunteers; morning surge; Amlodipine Besylate
MeSH Terms: conditions — Hypertension | interventions — Amlodipine

STUDY DESIGN:
Intervention Model Description: Test preparation (T): amlodipine besylate controlled-release tablets Specification: 5 mg Batch No.: 22102501 Content: 100.9% Expiry date: October 24, 2024 Storage conditions: dark, sealed at room temperature. Manufacturer: Overseas Pharmaceuticals, Ltd. Provider: Overseas Pharmaceuticals, Ltd.
  Reference preparation (R): amlodipine besylate tablets (trade name: Norfloxacin ®） Specification: 5 mg Batch No.: FX3445 Content: 100.2% Expiry date: January 2027 Storage conditions: dark and sealed Manufacturer: Pfizer Inc. Provider: Overseas Pharmaceuticals, Ltd.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Amlodipine besylate controlled-release tablets (Experimental): Test preparation (T): amlodipine besylate controlled-release tablets Specification: 5 mg Batch No.: 22102501 Content: 100.9% Expiry date: October 24, 2024 Storage conditions: dark, sealed at room temperature. Manufacturer: Overseas Pharmaceuticals, Ltd. Provider: Overseas Pharmaceuticals, Ltd. Take one tablet once a day.
  Interventions: Drug: Amlodipine besylate controlled-release tablets
- Amlodipine besylate tablets (trade name: Norfloxacin ®） (Active Comparator): Specification: 5 mg Batch No.: FX3445 Content: 100.2% Expiry date: January 2027 Storage conditions: dark and sealed Manufacturer: Pfizer Inc. Provider: Overseas Pharmaceuticals, Ltd. Take one tablet once a day.
  Interventions: Drug: Amlodipine besylate tablets (trade name: Norfloxacin ®）

INTERVENTIONS:
Drug: Amlodipine besylate tablets (trade name: Norfloxacin ®） — Specification: 5 mg Batch No.: FX3445 Content: 100.2% Expiry date: January 2027 Storage conditions: dark and sealed Manufacturer: Pfizer Inc. Provider: Overseas Pharmaceuticals, Ltd. Take one tablet once a day.
  Arms: Amlodipine besylate tablets (trade name: Norfloxacin ®）
Drug: Amlodipine besylate controlled-release tablets — Test preparation (T): amlodipine besylate controlled-release tablets Specification: 5 mg Batch No.: 22102501 Content: 100.9% Expiry date: October 24, 2024 Storage conditions: dark, sealed at room temperature. Manufacturer: Overseas Pharmaceuticals, Ltd. Provider: Overseas Pharmaceuticals, Ltd. Take one tablet once a day.
  Arms: Amlodipine besylate controlled-release tablets

SUMMARY:
Amlodipine Besylate Controlled-release Tablets in Healthy Volunteers in a Randomized, Open, Two-cycle, Double-cross, Fasting State Comparative Pharmacokinetic Study.

Major objective:

Taking amlodipine besylate controlled-release tablets (specification: 5 mg) developed by Overseas Pharmaceuticals, Ltd. as the test preparation and amlodipine besylate tablets (trade name: Luohuoxi, specification: 5 mg) produced by Pfizer Inc. as the control preparation, the pharmacokinetics parameters of the single oral administration test preparation and the control preparation in China healthy volunteers were investigated and compared in an fasting state.

Secondary objective:

To evaluate the safety of single oral administration of test preparation and control preparation in China healthy volunteers on an empty stomach.

DETAILED DESCRIPTION:
A single-center, randomized, open, two-cycle, double-cross, fasting experimental design method was adopted. All subjects must sign an informed consent form before taking part in the trial. Physical examination was conducted from the 14th day to the 1st day after administration, and the subjects the investigatorsre randomly assigned to one of the two sequential groups (T-R group and R-T group) according to the ratio of 1:1. That is, in the first cycle, 8 subjects in group T took one tablet of test preparation (amlodipine besylate controlled-release tablet, specification: 5mg) orally on an empty stomach; Group r: 8 subjects took one tablet of control preparation (amlodipine besylate tablet, Luohuoxi, specification: 5 mg) orally on an empty stomach, and about 240 ml of warm water was taken. Cross administration after 14 days.

On the morning of taking medicine, after the collection of blank blood samples, group T took one tablet of the test preparation (amlodipine besylate controlled-release tablets) orally; In group R, the oral control preparation (amlodipine besylate tablet) was taken with about 240 ml warm water. After 4 hours of administration, the standard meal was taken uniformly. Drinking water (except 240 ml water for medicinal purposes) is prohibited within 1 h before and 1 h after administration, and a unified diet is required during the experiment. The cleaning period was 14 days, and after 14 days, the drugs the investigatorsre administered in a cross way.

PK blood collection and blood sample treatment: 0 h before administration (within 1.0 h before administration) and 1.0 h, 2.0 h、3.0 h、3.5 h、4.0 h、4.5 h、5.0 h、5.5 h、6.0 h、6.5 h、7.0 h、7.5 h、8.0 h、8.5 h、9.0 h、10.0 h、12.0 h、14.0 h、16.0 h、24.0 h、36.0 h、48.0 h、72.0 h、96.0 h、144.0 h、168.0 h, a total of 27 time points to collect upper limb venous blood.

0 h before administration (within 1.0 h before administration) and 6.0± 0.5 h、12.0± 0.5 h、24.0±1.0 h、48.0±1.0 h、72.0±1.0 h、96.0±1.0 h、144.0±1.0 h、168.0±1.0 h after administration. The operating procedure of the second cycle is the same as that of the first cycle. In the second cycle, on the day after the sampling, the subjects need physical examination, vital signs examination, electrocardiogram and laboratory examination.

During the study, the investigators should observe and ask the subjective feelings of the subjects and the possible adverse reactions and events during the experiment. If the subject has AE during the trial, the researcher should try to follow up until the adverse events are relieved, or return to the screening level, or the subject's condition is stable.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects fully understand the purpose, nature, method and possible adverse reactions of the trial, voluntarily serve as subjects, and sign an informed consent form before any research procedure.
2. Healthy subjects over the age of 18 (including the age of 18) can be both male and female.
3. Male weight ≥ 50.0 kg, female weight ≥ 45.0 kg; Body mass index (BMI) is in the range of 19.0~26.0 kg/m2 (including the critical value).
4. From the signing of the informed consent form to the end of the study, there was no birth plan and voluntary adoption of appropriate and effective contraceptive measures, and there was no sperm or egg donation plan.
5. Subjects who can communicate well with researchers and understand and comply with the requirements of this study

Exclusion Criteria:

1. Allergic constitution, or a history of food or drug allergy or other allergic diseases (asthma, urticaria, eczema dermatitis, etc.); Or allergic to any component of amlodipine besylate.
2. Have a history of hypotension, or have a history of aortic stenosis or coronary artery occlusion.
3. Those who have poor condition of blood vessel puncture, or can not tolerate vein puncture, or have a history of needle and blood sickness.
4. There are cardiovascular, blood, liver, kidney, endocrine, respiratory, digestive, nervous, mental, immune, skin and metabolic disorders and other system diseases that researchers think are clinically significant, or there is a chronic or serious history of these diseases; Or there is a history of surgery that may affect drug absorption and metabolism.
5. Those with abnormal physical examination, vital sign examination, 12 lead ECG and laboratory examination, and those with clinical significance judged by the research doctor.
6. Human immunodeficiency virus (HIV) antibody, or hepatitis B virus surface antigen (HBsAg), or hepatitis C virus (HCV) antibody, or Treponema pallidum antibody (Anti TP) test results are positive.
7. Pregnant women, lactating women, or women of childbearing age have unprotected sexual behavior within 14 days before the planned administration, or the pregnancy test results are positive.
8. Those vaccinated within 3 months before screening (except for COVID-19 vaccine), or those vaccinated with COVID-19 vaccine within 1 week before screening, or those who plan to vaccinate any vaccine during the trial or within 1 week after the end of the study;
9. Or blood donation/blood loss ≥ 400 mL or blood transfusion or use of blood products within 3 months before screening, or blood donation (including blood components) planned during the test or within 3 months after the test.

   Previous medication:
10. Those who have a history of drug abuse or are positive for drug screening and have used drugs 6 months before screening, including MDMA (ecstasy), methamphetamine (methamphetamine), ketamine, morphine, tetrahydrocannabinol acid (cannabis).
11. Drugs that inhibit or induce liver metabolism of drugs (such as inducers: barbiturates, carbamazepine, phenytoin, glucocorticoids, omeprazole; inhibitors - SSRI antidepressants, cimetidine, diltiazem, macrolides, nitroimidazoles, sedatives and hypnotics, verapamil, fluoroquinolones, antihistamines, etc.) were used within 30 days before the first administration; Or 14 days before administration, any other drugs including prescription drugs, over-the-counter drugs, functional vitamins, health products or Chinese herbal medicine were used.

    Eating, smoking and drinking:
12. People with dysphagia, or those who have special requirements for diet and cannot accept a unified diet.
13. Those who used to drink too much caffeinated food or drink (such as coffee, strong tea, cola, chocolate, etc.) for a long time (more than 8 cups a day, 1 cup=250 mL), or take caffeinated food or drink within 72 hours before taking the drug for the first time, or can not be interrupted during the test.
14. Food rich in purine (such as anchovies, sardine, cow liver, cow kidney, etc.), or grapefruit products are eaten within 48 hours before administration, or cannot be interrupted during the test.
15. Those who have started significantly abnormal diet (such as diet and low sodium) within 4 weeks before screening.
16. Excessive smoking within 6 months before screening (average ≥ 5 cigarettes/day) or smoking within 48 hours before the first drug administration, or unable to stop using any tobacco products during the test period.
17. People who have a history of alcoholism or regularly drank alcohol within 6 months before screening, that is, people who drink more than 14 units of alcohol every week (1 unit=360 mL of beer with an alcohol content of 5%, 45 mL of spirits with an alcohol content of 40%, or 150 mL of wine with an alcohol content of 12%), or people who drink or eat food or drink containing alcohol within 48 hours before taking drugs for the first time, or people who have positive alcohol breath test on the day of their first stay, or who cannot stop drinking alcohol during the study period.

    other:
18. Those who have participated in or are participating in clinical trials of other drugs within 3 months before screening (defined as those who have used clinical research drugs).
19. Subjects who are judged by the investigator to be unsuitable for other factors in this clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2023-01-28 (Estimated); Primary Completion 2023-02-28 (Estimated); Study Completion 2023-03-10 (Estimated)

PRIMARY OUTCOMES:
Area under the curve from time zero to the time of the last quantifiable plasma | 1 month
  The 90% CI for the geometric mean ratios (i.e., antilog-transformation for 90% CI of difference with log transformation) of AUC0-last within [0.8, 1.25] range will be used to determine the result of bioequivalence.
Area under the curve from time zero to infinity (AUC0-inf) | 1 month
  The 90% CI for the geometric mean ratios (i.e., antilog-transformation for 90% CI of difference with log transformation)of AUC0-inf within [0.8, 1.25] range will be used to determine the result of bioequivalence.
Peak concentration at each treatment period (Cmax,tp) | 1 month
  The 90% CI for the geometric mean ratios (i.e., antilog-transformation for 90% CI of difference with log transformation)of Cmax,tp within [0.8, 1.25] range will be used to determine the result of bioequivalence.

SECONDARY OUTCOMES:
Peak concentration of the first dosing (Cmax) | 1 month
  Individual felodipine plasma concentration-time profile for each treatment period will be established.
Time to reach peak concentration of the first dosing (Tmax) | 1 month
  Individual felodipine plasma concentration-time profile for each treatment period will be established.
Terminal half-life (T1/2) | 1 month
  Individual felodipine plasma concentration-time profile for each treatment period will be established.
Mean residence time (MRT) | 1 month
  Individual felodipine plasma concentration-time profile for each treatment period will be established.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhujiang Hospital of Southern Medical University, Guangdong, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No